CLINICAL TRIAL: NCT00369603
Title: Functional Neuroimaging (fMRI) Biomarker of Allosteric Nicotinic Receptor Modulation in Mild Alzheimer's Disease Patients: A Razadyne vs. Aricept Dose Escalation Trial
Brief Title: Functional Brain Imaging of Medication Treatment Response in Mild Alzheimer's Disease Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Reduced access to AchEI medication-naive mild AD patients.
Sponsor: Duke University (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00011149; GAL-EMR-4026 (Other: DUMC)
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2008-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; fMRI; Functional Neuroimaging; Allosteric Nicotinic Receptor Modulation; Acetylcholinesterase Inhibition; Head to head; Dose escalation; Biomarker
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Razadyne ER (Experimental): galantamine treatment group
  Interventions: Drug: Razadyne ER
- Aricept (Experimental): Aricept Treatment Group
  Interventions: Drug: Aricept

INTERVENTIONS:
Drug: Razadyne ER — 4-weeks 8mg. Razadyne ER, then 4-weeks 16mg. Razadyne ER, and a subsequent 4-weeks of 24mg. Razadyne ER
  Arms: Razadyne ER
Drug: Aricept — 8-weeks 5mg. Aricept and a subsequent 4-weeks of 10mg. Aricept
  Arms: Aricept

SUMMARY:
The purpose of this study is to determine whether standard medications approved for Alzheimer's disease treatment differ in their action on brain functioning and whether any observed brain activity differences as result of treatment are associated with particular patterns of dementia improvement or reduced decline.

DETAILED DESCRIPTION:
This study seeks to differentiate task-related and resting brain activity patterns captured via functional magnetic resonance imaging (fMRI) and associated with two common Alzheimer's disease (AD) medications, equivalent in acetylcholinesterase inhibition effect (AChEI) but differing with respect to allosteric nicotinic receptor modulation effect. It is the primary aim of this project to gain a better understanding of the brain mechanisms involved in the attentional and executive skills improvements associated with nicotinic receptor modulation in mild AD patients.

To address this question, this 12-week continuous treatment, double-blind, head-to-head dose-escalation treatment trial seeks to visualize any treatment response unique to allosteric nicotinic receptor modulation and to associate these fMRI data with standard cognitive assessment outcomes. Using in-scanner tasks shown to reliably elicit brain activity in cortical regions important to memory and attention, this treatment trial will examine both resting and task-related BOLD signal characteristics in a well-characterized sample of 36 mild AD patients after periods of low dose and high dose AD dementia treatment with either galantamine hydrobromide (AChEI + nicotinic receptor modulation) or donepezil hydrochloride (AChEI only). Both the low and high dose imaging comparisons between treatment groups will be equivalent for 35% AChEI-effect, which may allow for the isolation of BOLD signal unique to allosteric nicotinic receptor modulation in both brain at rest and task-related brain states.

ELIGIBILITY:
Inclusion Criteria:

* Must meet diagnosis of mild Alzheimer's disease
* Must have a family member or caregiver who is willing to attend all study visits and provide information on your participation in the study
* If female, must be post-menopausal
* Must be able to swallow tablets

Exclusion Criteria:

* Metal implants or medical devises unsafe for MRI use
* Pre-menopausal female
* HIstory of recent head injury
* Significant major, life-threatening illness or injury (e.g., stroke, AIDS, etc.)
* Vascular dementia or any dementia other than Alzheimer's Disease
* History of significant alcoholism or drug abuse
* History of seizure disorder, developmental delay or major psychiatric illness

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Brain activity patterns, as collected via functional magnetic resonance imaging (fMRI), at rest and associated with task performance after 4 weeks of low-dose treatment and after 8-weeks of higher-dose treatment. | 4-weeks and 12-weeks

SECONDARY OUTCOMES:
Differences in cognitive testing and functional status at pre-treatment baseline and after completion of the 12-week treatment trial. | baseline and 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N Browndyke, PhD, Principal Investigator — Duke University; Roberto Cabeza, PhD, Principal Investigator — Duke University; James R Burke, PhD, Principal Investigator — Duke University; Kathleen Welsh-Bohmer, PhD, Principal Investigator — Duke University
Locations (1):
- Joseph & Kathleen Bryan Alzheimer's Disease Research Unit, Durham, North Carolina, United States